CLINICAL TRIAL: NCT02057198
Title: Exploratory Study of Impact of Oral Metronidazole, Vancomycin and Fidaxomicin on the Extent and Quantity of Host Carriage and Environmental Contamination With C. Difficile
Brief Title: Impact of Oral Antibiotic Treatment on C. Difficile
Acronym: C-Diff
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00043361
Record Dates: First submitted 2014-01-07; First posted 2014-02-06 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: C. Difficile; Diarrhea; Enterocolitis
MeSH Terms: conditions — Diarrhea; Enterocolitis | interventions — Fidaxomicin; Metronidazole; Benchmarking; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fidaxomicin (Active Comparator): 200 mg. 2 times a day for 10 days
  Interventions: Drug: Fidaxomicin
- Metronidazole (Active Comparator): 500 mg.orally 3 times daily for 10 days
  Interventions: Drug: Metronidazole
- Vancomycin (Active Comparator): 125 mg. orally 4 times a day for 10 days
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Fidaxomicin
  Other Names: Drug class(es): macrolides; Dificid
  Arms: Fidaxomicin
Drug: Metronidazole
  Other Names: Drug class(es): amebicides; Flagyl; Flagyl IV; Metro; Flagyl ER
  Arms: Metronidazole
Drug: Vancomycin
  Other Names: Drug Class:Glycopeptide antibiotics; Vancocin HCl Pulvules; Vancocin; Lyphocin; Vancocin HCl
  Arms: Vancomycin

SUMMARY:
The overall aim is to characterize and to compare the extent and quantity of C. difficile stool shedding, perianal colonization and environmental contamination in patients who received oral fidaxomicin, oral metronidazole, or oral vancomycin. This is a prospective, randomized, microbiologic and molecular, study of environmental contamination from patients with proven C. difficile associated diarrhea (CDAD).

DETAILED DESCRIPTION:
Background and Significance:

C. difficile has emerged as one of the most important pathogens that threaten the health and quality of life for many populations. Data from different studies clearly indicate that shedding of viable spores and subsequent contamination of environmental surfaces play an important role in the transmission of C. difficile. We aim to perform an analysis of the impact of different oral antibiotic therapy on microbiologic kinetics in patients with C. difficile diarrhea, such as: shedding, colonization and environmental contamination. We believe data from this study can inform whether drug therapies may be used to interrupt disease transmission and to improve the infection control of C. difficile.

Purpose of the Study:

The purposes of this study are to 1) determine the impact of oral fidaxomicin, oral metronidazole and oral vancomycin on the baseline and the temporal variation of C. difficile isolated from specific body sites of a patient with microbiology-proven CDAD and 2) determine the impact of oral fidaxomicin, oral metronidazole and oral vancomycin on the baseline and the temporal variation of C. difficile isolated from targeted surfaces in a hospital room. , More specifically, we will establish the extent and quantity of C. difficile shedding, colonization and environmental contamination in patients who received oral fidaxomicin, oral metronidazole, or vancomycin and the duration that stool remains positive for C. difficile.

This study will prospectively study the role of the environment in Healthcare Associated Infections (HAIs) in the modern healthcare setting and will specifically address many limitations of previous studies. The study will use modern diagnostic and molecular methods to describe the microbiologic characteristics and concordance of cultures from the environment and from patient, describe temporal variation and relationship in the microbiologic profiles of cultures obtained from the environment and from the patient, assess confounders such as hand hygiene and quality of cleaning, and provide longitudinal follow up for subsequent outcomes.

This study will utilize microbiologic and molecular techniques to critically and prospectively examine the impact of the environmental bioburden on the risk of colonization and infection of hospitalized patients. Data from this study will provide novel, important information regarding the true impact of the hospital environment on the acquisition and spread of HAIs and Multi-Drug Resistant (MDR)-pathogens in hospitalized patients over time. As such, data collected in this study may provide important information about the mechanisms and relative frequency of how and when environmental sources of bacteria lead to colonization and infection in hospitalized patients. These data may in turn stimulate or justify the future development of novel preventive interventions.

Design and Procedures/Study Interventions:

This is a randomized, controlled study of patients with documented CDAD, defined as having polymerase chain reaction for C. difficile in a patient with more than 3 loose stools within 24 hours. Eligible patients for enrollment will be identified by microbiology-driven alerts or by orders for contact isolation for C. difficile. Study team will be alerted to approach the patient to provide information about the study and to obtain informed consent.

This study will obtain microbiological cultures from 2 sources: 1) environmental surfaces in the room and 2) body surfaces of the patient at predefined intervals starting the day of enrol1ment. Cultures will be obtained on Day 1 (day of enrol1ment), Day 3 and Day 7 following admission to the room, at the end of each subsequent week (Day 14, Day 21, etc.), and on the day of discharge from the hospital room. Microbiological cultures will be obtained from the following body sites: perianal and stool specimens. Microbiological cultures will be obtained from 5 high-touch environmental surfaces as outlined in the protocol.

Selection of Subjects:

A total of 30 patients are anticipated to be enrolled in this study, 10 in each of the three treatment arms. Patients will be block-randomized to receive one of the three antibiotic treatments for CDAD described above. The study will enroll 10 patients receiving metronidazole therapy, 10 patients receiving oral vancomycin therapy and 10 patients receiving oral fidaxomicin therapy.

As soon as the PI or study coordinator finds that a patient has a positive C. difficile result, the primary care provider (PCP) in hospital will be contacted to discuss the patient. If the PCP agrees to allow potential enrollment, the PCP will introduce the study to the patient. If the patient indicates willingness to participate, the PI or study coordinator will be introduced by the PCP or another caregiver known to the patient. The informed consent process will take place if the patient is interested in participating. The patient will be enrolled as a study subject if all eligibility criteria are met. The PCP will formally prescribe fidaxomicin, metronidazole or vancomycin following randomization. Fidaxomicin will be supplied by the study sponsor. Metronidazole and vancomycin will not be supplied by the sponsor. If the subject is randomized to receive fidaxomicin, the PI or study coordinator will notify the Duke Investigational Drug Service (IDS) that a subject is enrolling and will order this drug through the IDS. As soon as the 10th subject who is prescribed fidaxomicin enrolls, then enrollment will be closed to patients prescribed fidaxomicin. Enrollment will be closed to subjects taking metronidazole and vancomycin as soon as the 10th subject in each group is enrolled. The subject will begin treatment with the medication prescribed by the PCP in hospital.

No compensation is being offered for participation in this study.

Consent Process:

The consent process will be conducted by a study coordinator or the principal investigator. This will typically occur in the patient's hospital room..

Subject's Capacity to Give Legally Effective Consent:

Subjects will need to be able to give consent to participate in this study.

Risk/Benefit Assessment:

The risks are minimal for this study. First, patients may experience adverse effects from the antibiotics that they consent to receive. Each of three agents is recommended for the treatment of CDAD. Second, the microbiological samples that will be taken may cause some discomfort and minor bleeding which will be discussed with the patient during the consenting process. Declining to participate in the study will not affect the clinical care of the patient. Results of study specimens will not be analyzed in real-time and will not be sent back to clinicians.

SAEs are not anticipated for this study. Any standard SAE events that may occur will be reported to the manufacturer and to the IRB.

There is no direct benefit to the patient in the study. The sponsor will supply Fidaxomicin if this is prescribed for a patient enrolled in the study. The data from this study may prompt future studies that examine the use oral antibiotics to reduce the transmissibility of C. difficile.

Data Analysis and Statistical Considerations:

Descriptive statistics will be used to correlate culture results from the environment and the patient.

Data and Safety Monitoring:

PI will review and sign off on all adverse events or problems as they occur and will submit reports of such events to the IRB in accordance with HRPP policies and to the sponsor in accordance with the protocol.

Privacy, Data Storage and Confidentiality:

Privacy during swabbing shall be maintained by swabbing the patient in the patient's room with the door closed as would be appropriate for other patient care, using Universal Precautions. To ensure privacy the patient and environmental samples will use an automatically generated ID and room number in place of name, MRN or other personal identifiers.

Data collected by the study will be entered into secure Access databases. All connections to the system, both external and internal, occur over encrypted channels. Access to components of the system is role-based and can only be granted by administrators of the system. All collected information is stored on a server hosted by Duke Medicine.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with microbiology-proven CDAD
* provides informed consent
* eligible to receive oral antibiotic therapy

Exclusion Criteria:

* prisoners
* pregnant women
* children <18 years
* patients who have contra-indications for perianal swabs, those who has medical conditions that would invalidate the results of the swabs
* patients requiring intravenous therapy for treatment of CDAD
* patients who do not consent and those who withdraw consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-06-10 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Sexton, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Turner NA, Warren BG, Gergen-Teague MF, Addison RM, Addison B, Rutala WA, Weber DJ, Sexton DJ, Anderson DJ. Impact of Oral Metronidazole, Vancomycin, and Fidaxomicin on Host Shedding and Environmental Contamination With Clostridioides difficile. Clin Infect Dis. 2022 Mar 1;74(4):648-656. doi: 10.1093/cid/ciab473. PMID 34017999

RESULTS

PARTICIPANT FLOW:
Groups:
- Fidaxomicin: 200 mg. 2 times a day for 10 days
  Fidaxomicin
- Metronidazole: 500 mg.orally 3 times daily for 10 days
  Metronidazole
- Vancomycin: 125 mg. orally 4 times a day for 10 days
  Vancomycin
Period: Overall Study
Arm/Group | Fidaxomicin | Metronidazole | Vancomycin
Started | 11 | 11 | 11
Completed | 11 | 10 | 10
Not Completed | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Discharged early; lost to followup | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only participants who completed the study are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fidaxomicin | Metronidazole | Vancomycin | Total
Number analyzed (Participants) | 11 | 10 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (22) | 62.2 (15.1) | 63.4 (9.6) | 62 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 5 | 15
  Male | 7 | 4 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 10 | 10 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 4 | 14
  White | 6 | 5 | 6 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Median Total Colony Forming Units (CFU) of C. Difficile Identified in the Hospital Room Environment for Each Antibiotic Treatment Group.
Description: Rodac plates were used to take environmental samples from 5 different sites within each patient's hospital room (bedrail, overbed table, sink, toilet seat, bathroom floor). Each Rodac plate samples a surface area of ~25 cm2. 5 replicates were taken for each site and repeated on days 0, 3, 7, and 14. Median total colony counts are reported for each treatment group. Data from the specified time points were combined to construct a decay slope, representing the reduction in log(CFUs)/day for each treatment group. We compared the slope (rate of change) between treatment groups using mixed effects models.
Time Frame: Days 0, 3, 7 and 14.
Population: Only completed participants were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: Colony forming units (CFUs)
Arm/Group | Fidaxomicin | Metronidazole | Vancomycin
Number analyzed (Participants) | 11 | 10 | 10
Colony forming units (CFUs)
  Day 0 | 56 [0 to 158] | 33 [23 to 43] | 149 [0 to 227]
  Day 3 | 7 [4 to 9] | 53 [17 to 92] | 24 [5 to 43]
  Day 7 | 0 [0 to 0] | 15 [12 to 18] | 0 [0 to 0]
  Day 14 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Metronidazole vs Vancomycin; Test type: Superiority; p = 0.52, Mixed Models Analysis — Data from the specified time points were combined to construct a decay slope, representing the reduction in log(CFUs)/day for each treatment group. We compared the slope (rate of change) between treatment groups using mixed effects models; A mixed effects model was used to compare decay slopes for the reduction in log(CFUs)/day according to each treatment group; Slope = -0.15, 95% CI 2-sided [-0.34 to 0.05]
Statistical Analysis 2: Comparison: Fidaxomicin vs Metronidazole; Test type: Superiority; p = 0.66, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Slope = -0.17, 95% CI 2-sided [-0.69 to 0.35]

2. Secondary Outcome: Total Environmental Contamination According to Antibiotic Treatment Group
Description: In addition to total colony counts over time, the investigators also assessed the proportion of positive cultures over time (from the 5 replicate Rodac plate samplings repeated at each of 5 sites within each patient room: bedrail, overbed table, sink, toilet seat and bathroom floor). The cumulative proportion of positive cultures (including days 0, 3, 7, 14) is reported according to each treatment group.
Time Frame: Days 0, 3, 7, and 14
Population: Only completed participants were included in the analysis.
Measure: Number; unit: percentage of positive cultures
Units Other Than Participants: Environmental cultures
Arm/Group | Fidaxomicin | Metronidazole | Vancomycin
Number analyzed (Participants) | 11 | 10 | 10
Number analyzed (Environmental cultures) | 794 | 575 | 774
percentage of positive cultures | 13.4 | 18.6 | 7.6
Statistical Analysis 1: Comparison: Metronidazole vs Vancomycin; Test type: Superiority; p < 0.001, Chi square (2 proportion test)
Statistical Analysis 2: Comparison: Fidaxomicin vs Metronidazole; Test type: Superiority; p = 0.01, Chi square (2 proportion test)

3. Secondary Outcome: Molecular Relatedness of Isolates
Description: When sufficient growth was available to permit sub-culture and ribotyping, we conducted ribotyping of each patient's stool C. difficile isolate for comparison to isolates from the same patient's hospital environment. Reported is the total percent of hospital room environmental isolates that match the ribotyping of the associated patient's stool sample (there is no averaging).
Time Frame: Days 0-14
Population: Ribotyping could only be conducted in instances where sufficient growth occurred from both patient and environmental samples to permit subculture.
Measure: Number; unit: percent of matching isolates
Units Other Than Participants: Environmental Isolates
Arm/Group | Fidaxomicin | Metronidazole | Vancomycin
Number analyzed (Participants) | 3 | 4 | 4
Number analyzed (Environmental Isolates) | 22 | 25 | 9
percent of matching isolates | 68.1 | 80.0 | 77.8
Statistical Analysis 1: Comparison: Metronidazole vs Vancomycin; Test type: Superiority; p = 0.99, Chi square (2 proportion test)
Statistical Analysis 2: Comparison: Fidaxomicin vs Metronidazole; Test type: Superiority; p = 0.52, Chi square (2 proportion test)

4. Secondary Outcome: C. Difficile Shedding in Stool Over Time
Description: C. difficile was isolated and serially diluted to permit colony counts (CFU/g stool) over time for each patient.
Time Frame: Days 0, 3, 7, 14
Population: Only completed participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: CFU/g stool
Arm/Group | Fidaxomicin | Metronidazole | Vancomycin
Number analyzed (Participants) | 11 | 10 | 10
CFU/g stool
  Day 0 | 815940 (949503) | 2233564 (3845558) | 35340 (41612)
  Day 3 | 72200 (156429) | 1200 (283) | 400 (693)
  Day 7 | 0 (0) | 0 (0) | 0 (0)
  Day 14 | 0 (0) | 0 (0) | 0 (0)
Statistical Analysis 1: Comparison: Metronidazole vs Vancomycin; Data from the specified time points were combined to construct a decay slope, representing the reduction in log(CFUs)/day for each treatment group. We compared the slope (rate of change) between treatment groups using mixed effects models. Data from the specified time points were combined to construct a decay slope, representing the reduction in log(CFUs)/day for each treatment group. We compared the slope (rate of change) between treatment groups using mixed effects models; Test type: Superiority; p = 0.05, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Slope = -0.43, 95% CI 2-sided [-0.67 to -0.19]
Statistical Analysis 2: Comparison: Fidaxomicin vs Metronidazole; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Slope = -0.85, 95% CI 2-sided [-1.14 to -0.57]

5. Secondary Outcome: Count of Stool Specimens From Patients That Are Positive for C. Difficile
Description: Count of stool cultures positive for C. difficile at each time point
Time Frame: Days 0, 3, 7, 14
Population: Only completed participants were included in the analysis.
Measure: Number; unit: Number of positive stool cultures
Units Other Than Participants: specimens
Arm/Group | Fidaxomicin | Metronidazole | Vancomycin
Number analyzed (Participants) | 11 | 10 | 10
Number analyzed (specimens) | 20 | 22 | 20
Number of positive stool cultures
  Day 0 | 20 | 21 | 17
  Day 3: number analyzed (specimens) | 10 | 4 | 6
  Day 3 | 6 | 3 | 2
  Day 7: number analyzed (specimens) | 4 | 2 | 4
  Day 7 | 0 | 0 | 0
  Day 14: number analyzed (specimens) | 2 | 2 | 4
  Day 14 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Stool Specimens From Patients That Are Positive for C. Difficile
Description: Percentage of stool cultures positive for C. difficile at each time point
Time Frame: Days 0, 3, 7, 14
Population: Only completed participants were included in the analysis.
Measure: Number; unit: % of positive stool cultures
Units Other Than Participants: specimens
Arm/Group | Fidaxomicin | Metronidazole | Vancomycin
Number analyzed (Participants) | 11 | 10 | 10
Number analyzed (specimens) | 20 | 22 | 20
% of positive stool cultures
  Day 0 | 100 | 95.5 | 85
  Day 3: number analyzed (specimens) | 10 | 4 | 6
  Day 3 | 60 | 75 | 33
  Day 7: number analyzed (specimens) | 4 | 2 | 4
  Day 7 | 0 | 0 | 0
  Day 14: number analyzed (specimens) | 2 | 2 | 4
  Day 14 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Metronidazole vs Vancomycin; Test type: Superiority; p = 0.48, Chi square (two proportion test)
Statistical Analysis 2: Comparison: Fidaxomicin vs Metronidazole; Test type: Superiority; p = 0.66, Chi square (two proportion test)

ADVERSE EVENTS:
Time Frame: During of index hospital admission (estimated maximum of 4 weeks after enrollment).
Arm/Group | Fidaxomicin | Metronidazole | Vancomycin
All-Cause Mortality (participants affected / at risk) | 2/11 | 0/10 | 2/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT02057198/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT02057198/SAP_001.pdf